CLINICAL TRIAL: NCT00395785
Title: Protection During Carotid Stenting in High Risk Patients With the TriActiv ProGuard System
Brief Title: Evaluation of the TriActiv ProGuard System During Carotid Artery Stenting
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor elected to not pursue this indication for the study device.
Sponsor: Kensey Nash Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROGUARD
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Carotid Stenosis
Keywords: Carotid stenosis; Intracranial Embolism; Carotid artery; Carotid stent; Embolic protection; TriActiv ProGuard System; Carotid angioplasty
MeSH Terms: conditions — Carotid Stenosis; Intracranial Embolism | interventions — Embolic Protection Devices

INTERVENTIONS:
Device: Carotid Stent Implantation
Device: Embolic Protection

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the TriActiv® ProGuard™ System when used during a stent placement in a blockage within the carotid artery in patients considered to be at high risk for complications from surgical endarterectomy.

DETAILED DESCRIPTION:
Patients with certain anatomic or medical conditions have a greater risk of serious complications following carotid endarterectomy (a surgical procedure that removes blockages in the carotid artery). Recently, these patients have been treated effectively with the implantation of a carotid stent (a metallic mesh tube). When implanting the carotid stent, physicians use devices called embolic protection devices to prevent particles from the blockage from flowing up to the brain. The TriActiv® ProGuard™ System is an embolic protection device that uses a small balloon to temporarily stop blood flow within the diseased carotid artery while the stent is implanted. Then, the TriActiv® ProGuard™ System removes any particles that may have been released from the blockage during stent implantation before blood flow is restored. This study will evaluate the safety and efficacy of the TriActiv® ProGuard™ System during carotid stent placement in patients who are considered to be at a high risk for complications from surgical endarterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 year of age
* Patient gives informed consent
* Less than 30mm stenosis in the common and/or internal carotid artery: at least a 50% stenosis if symptomatic or at least an 80% stenosis if asymptomatic
* At least one medical or anatomic condition which makes the patient a high surgical risk.

Exclusion Criteria:

* Stroke within 14 days
* Major stroke with significant residual effects
* Myocardial infarction within 72 hours
* Extensive atherosclerotic disease in the aortic arch or proximal common carotid artery
* Severe carotid artery tortuosity
* Total occlusion
* Presence of thrombus or heavy calcification in the carotid artery
* Pre-existing carotid artery dissection
* Any planned interventional or surgical procedures within 30 days
* Atrial fibrillation
* Creatinine > 2 mg/dL
* Current participation in another investigational drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
A composite of major adverse events including any death, any stroke and/or myocardial infarction through thirty days post-procedure.

SECONDARY OUTCOMES:
Rate of subject intolerance to prolonged carotid artery occlusion;
Rate of access site complications requiring treatment with blood transfusion or surgical repair.
Rate of successful use of the study device success
Rate of successful lesion treatment
Rate of procedure success

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Roubin, MD, Principal Investigator — Lenox Hill Hospital, New York, NY; Rajesh Dave, MD, Principal Investigator — Pinnacle Health Hospital, Harrisburg, PA
Locations (34):
- United States (31):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Brotman Medical Center, Beverly Hills, California
  - Good Samaritan Hospital, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - Stanford University Medical Center, Stanford, California
  - Florida Crdiovascular Research at JFK Medical Center, Atlantis, Florida
  - University of Florida, Jacksonville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Mt. Sinai Medical Center, Miami Beach, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Crawford Long Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Jewish Hospital, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Millard Fillmore Hospital, Buffalo, New York
  - Millard Fillmore, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Lenox Hill Hospital, New York, New York
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Lorain Community Hospital, Elyria, Ohio
  - St. John West Shore Hospital, Westlake, Ohio
  - Pinnacle Health Hospital, Harrisburg, Pennsylvania
  - St. Joseph Medical Center, Wyomissing, Pennsylvania
  - Sisters of Charity Providence Hospital, Columbia, South Carolina
  - Methodist Germantown, Germantown, Tennessee
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - LDS Hospital, Salt Lake City, Utah
  - Virginia Cardiovascular Specialists/St. Mary's Hospital, Richmond, Virginia
- Germany (3):
  - Stadtisches Krankenhaus Neuperlach, Bayern
  - CardioVasculares Centrum Frankfurt Sankt Katharinen, Frankfurt
  - Herzzentrum Hamburg, Hamburg